CLINICAL TRIAL: NCT02748590
Title: Evaluation of Sacral Neuromodulation (SNM) in the Treatment of Active Ulcerative Colitis
Brief Title: Evaluation of Sacral Neuromodulation (SNM) in the Treatment of Active Ulcerative Colitis (PRIMICISTIM)
Acronym: PRIMICISTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0448
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Active Ulcerative Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuromodulation (Experimental)
  Interventions: Device: InterStim II Neurostimulator Model 3058

INTERVENTIONS:
Device: InterStim II Neurostimulator Model 3058 — The neuromodulation will be carried out according to the usual protocol: Hospitalization for the establishment of percutaneous electrode in the operating room under general anesthesia with fluoroscopic control. The pacemaker startup will be performed within 12h after surgery

SUMMARY:
Efficacy of ulcerative colitis to induce remission in patients with moderate to severe active ulcerative colitis.

DETAILED DESCRIPTION:
Neuromodulation is a validated option for the treatment of fecal incontinence. Safety of this original approach has been confirmed by several studies. New indications for this minimally-invasive procedure are actually under evaluation particularly in the fields of irritable bowel syndrome and chronic constipation with promising results. Its mechanism of action remains partially unknown and the target of neuromodulation is not limited to the anal sphincter but the whole colonic motility seems to be influenced by this therapeutic approach. Moreover, recent experimental studies have shown that neuromodulation was able to reinforce the intestinal epithelial barrier involved in the pathophysiology of ulcerative colitis.

Subsequently, preliminary results in human have shown improvement of inflammation in patients suffering from inflammatory bowel diseases. In fact, despite recent improvement in medical therapies in inflammatory bowel diseases and particularly in ulcerative colitis, several patients are suffering from disabling chronic active disease. In those cases of refractory diseases, the only alternative treatment is a pan-proctocolectomy and ileal pouch surgery. This approach is a curative option, but leads to a significant morbidity and frequent functional disorders in the long-term follow-up (permanent stoma in 7 to 10% of the cases). Moreover, in limited distal disease (left colon and rectum) the surgical option seems to be unadapted and many patients remain symptomatic and suffer chronic active disease.

The aim of this study will be to assess in a prospective pilot study the efficacy of ulcerative colitis in inducing the remission of chronic active ulcerative colitis limited to the left side of the colon and improving the quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Active Ulcerative Colitis diagnosed on criteria Lennard Jones (31) for at least 1 year
* > 18 yo
* E1 - E2 disease or extended to transverse colon but not beyond the hepatic flexure (endoscopic pictures)
* resistant to medical treatment: active after introduction for at least 8 weeks of maintenance treatment (immunosuppressive or anti-TNF)
* Activity score >5 and endoscopic score >2
* Absence of bacterial infection in progress (Clostridium difficile)
* Affiliated with a social protection scheme and had signed an informed consent

Exclusion Criteria:

* Severe forms requiring hospitalization an intravenous treatment or immediate surgery
* infectious colitis or proctitis
* Prednisone> 20 mg / d
* Contraindications to the use of neuromodulator
* Corticosteroid therapy by intravenous route
* Pregnant women
* Major Trust

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of neuromodulation to induce remission at Week 8 in patients with moderate to severe active ulcerative colitis (Mayo score) | 8 weeks
  Clinical and endoscopic remission as measured by the Mayo score ≤ 2 points without any criteria> 1 point to week 8

SECONDARY OUTCOMES:
Assess the Remission at Week 16 ( Mayo score) | 16 weeks
  Remission is defined by a Mayo score ≤ 1 point.
Assess the Response at Week 8 and Week 16 (scale Ulcerative Colitis Disease Activity Index) | 16 weeks
  The response is defined as a decrease of at least 1 point in the item assessment by the physician and at least 1 point from the 3 other items with no increase in the other dimensions of the score.
Assess the clinical response at Week 8 and Week 16 (scale Ulcerative Colitis Disease Activity Index) | 16 weeks
  The answer Clinic is defined as a decrease of at least 3 points in the score Clinic dimension compared to baseline.
Assess the endoscopic response at Week 8 and Week 16 (scale Ulcerative Colitis Disease Activity Index) | 16 weeks
  Endoscopic response corresponds to a decrease of at least 1 point in the endoscopic score
Assess the histological response at Week 8 and Week 16 (Geboes Score) | 16 weeks
  Mucosal healing is defined by a score of Geboes less than or equal to 1 of the biopsy examination
Assess the biological response at Week 8 and Week 16 (C-reactive protein) | 16 weeks
  Biological response is defined as a decrease of C-reactive protein
Assess the biological response at Week 8 and Week 16 (Calprotectin) | 16 weeks
  Biological response is defined as a decrease of fecal calprotectin.
Evaluate the symptom's resolution at Week 3, Week 8 and Week 16 (scale Ulcerative Colitis Disease Activity Index) | 16 weeks
  The resolution is defined by bleeding Ulcerative Colitis Disease Activity Index sub-score 0
Evaluate the urgencies cessation at Week 3, Week 8 and Week 16 (scale Ulcerative Colitis Disease Activity Index) | 16 weeks
  The resolution is defined by bleeding Ulcerative Colitis Disease Activity Index sub-score 0
Evaluate the cessation of rectal bleeding at Week 8, Week 16 | 16 weeks
  Cessation of rectal bleeding is defined as rectal bleeding Ulcerative Colitis Disease Activity Index sub-score of 0
Evaluate the immunosuppressive drugs at Week 8 and Week 16 | 16 weeks
  Absence or decreasing in immunosuppressive drugs during the follow-up
Evaluate the need for steroids at Week 8 and Week 16 | 16 weeks
  The need for steroid treatment at least once during the follow-up period
Evaluate the tolerance of neuromodulation in Ulcerative Colitis patients at Week 3, Week 8 and Week 16 | 16 weeks
  Tolerance of neuromodulation is stated by symptom specific scale
Evaluate the quality of life of the patients at Week 8 and Week 16 (Scale The Short Form 36) | 16 weeks
  Quality of life is evaluated with The Short Form 36 scale
Assess abdominal discomfort for weeks at Week 8 and Week 16 | 16 weeks
  Bristol Stool Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France